CLINICAL TRIAL: NCT05589740
Title: Wellness With Culturally Optimized Messages for Ethnic-diverse Latinos
Brief Title: Culturally Optimized Messages for Latinos
Acronym: WELCOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Josiemer Mattei, Donald and Sue Pritzker Associate Professor of Nutrition, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB22-0828
Record Dates: First submitted 2022-10-14; First posted 2022-10-21 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Diet, Healthy; Diet Habit; Obesity; Blood Pressure; Psychological
MeSH Terms: conditions — Feeding Behavior; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group consisting of culturally-tailored healthy eating advice through daily text messages for 2 months (delivery phase); a subsequent reinforcement phase of 2-months to repeat the text messages; and a subsequent maintenance phase of 2-months with no text messages.
  Interventions: Behavioral: Culturally tailored healthy eating advice
- Control (Active Comparator): Control group consisting of general healthy eating advice through daily text messages for 2 months (delivery phase); a subsequent reinforcement phase of 2-months to repeat the text messages; and a subsequent maintenance phase of 2-months with no text messages.
  Interventions: Behavioral: Standard healthy eating advice

INTERVENTIONS:
Behavioral: Culturally tailored healthy eating advice — Culturally-tailored education includes strategies for healthy eating, preferences for traditional healthy foods, recommendations for limiting unhealthy traditional foods, portion sizes, etc.
  Arms: Intervention
Behavioral: Standard healthy eating advice — Standard healthy eating education includes strategies, foods, portions, and cooking and eating tips for general dietary recommendations from USDA My Plate
  Arms: Control

SUMMARY:
This project aims to redesign and optimize a deep-structure culturally-tailored healthy eating program and test its effectiveness in improving dietary outcomes, anthropometric, and blood pressure among 75 diverse Latinos, compared to surface-level messages.

DETAILED DESCRIPTION:
This project aims to redesign and optimize a deep-structure culturally-tailored healthy eating program and test its effectiveness in improving dietary outcomes, anthropometric, and blood pressure among 75 diverse Latinos, compared to surface-level messages. The WELCOME study will be based on the RE-AIM framework with improved reach, adoption, implementation, and maintenance strategies. The intervention arm is a deep-structure cultural tailored text messages for distinct Latino heritages (e.g., Caribbean and non-Caribbean) informed by mixed-methods formative research, compared to surface-level healthy eating messages based on the USDA My Plate Spanish version. The program runs for 6 months: 2-months delivery phase + 2-months reinforcement phase + 2-months maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

* age 25-65 y/o
* self-reported Hispanic/Latino heritage
* able to understand and answer questions in Spanish or English
* living in Massachusetts for the past year and not planning to move in the next year
* having a cellphone with the capacity of receiving and sending text messages and giving consent for the Study to text this number as part of the intervention

Exclusion Criteria:

1. self-reported diagnosis of cancer, diabetes or major stomach or heart condition (e.g.: gastrointestinal cancers, coronary heart disease, previous stroke or heart attack, severe dietary allergies or restrictions)
2. planning to move Massachusetts in the next year
3. currently pregnant
4. institutionalized (i.e.: hospital, prison, etc.).

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Changes in diet quality score | Month 4
  Determine the change in score of short diet quality screener (range 18-54; from lowest to highest quality)
Change in levels of adipose risk factor | Month 4
  Estimate the change in the value of waist circumference (cm)
Change in levels of blood pressure risk factor | Month 4
  Estimate the change in the value of systolic and diastolic blood pressure (mmHg)
Change in dietary habits | Month 4
  Determine the change in the score of dietary behaviors (range 1-5)

SECONDARY OUTCOMES:
Changes in diet satisfaction: diet satisfaction scale | Month 4
  Determine the change in the score of the Diet Satisfaction Questionnaire (DSat-45) (range 45-225; from lowest to highest satisfaction) and its summed seven subscales (ranges 5-40

CONTACTS AND LOCATIONS:
Overall Officials: Josiemer Mattei, PhD, Principal Investigator — Harvard Chan School of Public Health
Locations (1):
- Harvard TH Chan School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Study personnel will manage and distribute the data generated from the study with other investigators observing NIH policy on the dissemination and sharing of research results. Study information and requests for data will be available immediately upon the data being coded and properly revised for quality control after culmination of the study; deidentified data will be available upon request.

DOCUMENTS (1):
  • Informed Consent Form (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT05589740/ICF_000.pdf